CLINICAL TRIAL: NCT04119232
Title: A Randomized, Clinical Trial Evaluating Methods to Increase Physical Activity After a Pregnancy Complicated by a Hypertensive Disorder
Brief Title: Randomized Clinical Trial to Increase Physical Activity After a a Hypertensive Pregnancy
Acronym: STEPUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 833609
Record Dates: First submitted 2019-10-07; First posted 2019-10-08 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Hypertension in Pregnancy; Preeclampsia; Gestational Hypertension
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia

STUDY DESIGN:
Intervention Model Description: We will conduct a two-arm randomized, controlled trial comparing a control group that uses wearable devices to track physical activity to an intervention group that uses the same wearable devices and participates in a team-based model of social incentives that gamifies physical activity. Patients will be randomized to one of the two arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Individual participants will use a wearable device to monitor daily step counts, set a step goal, and receive automated daily feedback on step goal attainment.
- Social incentives-based program (Experimental): Individual participants will use a wearable device to monitor daily step counts, set a step goal, and receive automated daily feedback on step goal attainment. Participants will be placed on a team of 3 randomly assigned participants and receive the social incentives intervention.
  Interventions: Behavioral: Social incentives-based program

INTERVENTIONS:
Behavioral: Social incentives-based program — Individual participants will use a wearable device to monitor daily step counts, set a step goal, and receive automated daily feedback on step goal attainment. Participants will be placed on a team of 3 randomly assigned participants and receive the social incentives intervention.
  Arms: Social incentives-based program

SUMMARY:
STEPUP is a 12-week randomized clinical trial among 126 postpartum women with pregnancies complicated by hypertensive disorders. Participants will be randomized to a control arm and receive a Fitbit or an intervention arm. The intervention arm will receive a Fitbit and set a step count goal, receive daily feedback via text about whether they reached their goal, and will be placed in virtual teams with other participants where they can win points for their team if they meet their daily goals. The main study outcomes will be increase in mean step count and change in psychosocial survey measures.

DETAILED DESCRIPTION:
Women with hypertensive disorders of pregnancy, such as preeclampsia and gestational hypertension, are at elevated risk of developing hypertension, diabetes, heart failure, and premature atherosclerotic cardiovascular disease. Current guidelines recommend intensive lifestyle modification for women with a history of hypertensive disorders in pregnancy in order to reduce the risk of developing cardiometabolic risk factors or overt CV disease. However, limited research exists to guide how to implement lifestyle modification for this population. The postpartum period poses unique challenges to adopting a healthy lifestyle. Remote interventions using mobile technology may be particularly effective. Social incentives designed using insights from behavioral economics have been demonstrated to motivate health behavior change, such as increasing physical activity. The objective of this study is to use a randomized clinical trial to test the effectiveness of a 12-week team-based, mobile health interventions using wearable devices and social incentives to increase physical activity in the postpartum period.

ELIGIBILITY:
Inclusion Criteria:

* Delivered a live baby at HUP or PAH within 4.0-12.6 weeks prior to study enrollment;
* Diagnosis of chronic hypertension, gestational hypertension, or preeclampsia during most recent pregnancy;
* Participating in Heart Safe Motherhood (HSM) program;
* Ability to read and provide informed consent to participate in the study;
* Has smartphone and email address

Exclusion Criteria:

* Does not speak English
* Answers yes to any of the following questions:
* Are you currently participating in any other physical activity studies?
* Do you have any medical conditions or other reasons why you could not participate in a 12-week physical activity program?
* Participants will be excluded after completing the baseline period if their baseline step count is too high (greater than or equal to 10,000 steps per day).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
Change in mean daily steps | weeks 3 to 14 of the intervention
  Change in mean daily step count from the baseline period (weeks 1-2) to the intervention period (weeks 3-14)

SECONDARY OUTCOMES:
Proportion of participant-days that step goals are achieved | weeks 3 to 14 of the intervention
  proportion of days participants meet their step goal
Mean daily steps during the 12-week intervention period adjusted for baseline step count | 12-week intervention period
  Mean daily steps during the 12-week intervention period adjusted for baseline step count
Change in perceived social support scale | weeks 3 to 14 of the intervention
  As measured by the "multidimensional scale of perceived social support", MS-PSS -- a 12-item scale designed to measure perceived social support from three sources: Family, Friends, and a Significant Other. Scored 1-12, with 1 having the lowest support and 12 having high support.
Change in Edinburgh postnatal depression scale (EPDS) | weeks 3 to 14 of the intervention
  Change in Edinburgh postnatal depression scale (EPDS): scored 0-30 with a score of 10 or greater indicating depressive symptoms
Change in Systolic blood pressure | weeks 3 to 14 of the intervention
Change in Diastolic blood pressure | weeks 3 to 14 of the intervention
Change in weight | weeks 3 to 14 of the intervention
Change in hypertension diagnosis | weeks 3 to 14 of the intervention
Health care utilization (attended postpartum OB visit or postpartum visit with primary care or cardiology) | weeks 3 to 14 of the intervention
Change in breastfeeding rates | weeks 3 to 14 of the intervention
Change in sleep duration as measured by Fitbit | weeks 3 to 14 of the intervention
Moderate or vigorous activity, as measured by Fitbit | weeks 3 to 14 of the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No